CLINICAL TRIAL: NCT06184724
Title: Implementation Pilot of Preoperative CGA Referral Process for Older Patients Undergoing Major Surgery
Brief Title: Implementation Pilot of Preoperative CGA Before Major Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-1692; 1K23AG081487 (NIH); A539707 (Other: UW Madison)
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Surgery; Geriatric Assessment; Health Services Research; Implementation Science

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from surgery clinics in a pre-post trial. The comparison group is a historic baseline for routine care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post Implementation (Experimental): Participants will be recruited from surgery clinics in the post-implementation group. They will go through a streamlined referral process as part of an implementation package for CGA before surgery.
  The control group will be historic baseline data. That is, older surgical patients who were treated Pre-Implementation. These patients would have received standard, routine clinical care without the use of the implementation package.
  Interventions: Other: Implementation Package for CGA; Other: Routine Clinical Care

INTERVENTIONS:
Other: Implementation Package for CGA — The Implementation Package will include streamlined referral processes and education for surgeons and staff about the new processes. These strategies will be applied after surgery is ordered to help increase the reach and adoption of the CGA.
Other: Routine Clinical Care — Routine care may or may not include the use of the CGA before surgery. The use of CGA in clinical care is up to the medical and surgical healthcare providers.

SUMMARY:
The goal of this clinical trial is to test whether a new implementation package can help older adults prepare for major surgery. The main question it aims to answer is: Can the implementation package help give more people access to this resource? Participants will be in two groups: older adults who are planning a major surgery and their medical and surgical healthcare providers. The results will be compared to a historic baseline.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test a new implementation package, which will be applied at the clinic-level, to see whether it can help more older adults prepare for major surgery. The study will evaluate whether the implementation package (1) improves the number of older adults who get a full "comprehensive geriatric assessment" (CGA) before surgery compared to the number of older adults who would be eligible for it, also called "reach"; and (2) increases the use of CGA by the medical and surgical providers who are taking care of these older adults, also called "adoption".

Participants will be in two groups: older adults who are planning a major surgery and their medical and surgical healthcare providers. The implementation package will include streamlined referral processes and education for surgeons and staff about the new processes. The results will be compared to a historic baseline

Findings from this study will help the lead researcher design a larger trial that will test both the implementation (or how something is done) at the same time as it tests the effectiveness (how well it works).

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 80 or older who is scheduled for an elective inpatient major surgery
2. Provider working in a clinic where pCGA is performed or a related anesthesia pre-operative clinic
3. Surgeon with a patient aged 80 or older who is scheduled for an elective inpatient major surgery

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients referred divided by number of eligible patients | 6 and 12 months after implementation
  Reach to potentially eligible patients will be measured by the number of patients referred divided by number of eligible patients.
Number of surgeons placing referral orders divided by the number of surgeons | 6 and 12 months
  Adoption by Referring Surgeons will be measured by the number of surgeons placing referral orders divided by the number of surgeons

SECONDARY OUTCOMES:
Fidelity: Percent of completed CGA components per visit | 30 days after visit
  Fidelity of the intervention or degree to which the CGA is delivered as intended will be measured by the percent of completed CGA components per visit.
Feasibility of Intervention Measure (FIM) Score | 6 and 12 months
  Perceived ease of use of implementation package will be measured by the 4-item validated Feasibility of Intervention Measure. Mean scores between 1 and 5 will be reported, where higher scores increased feasibility.
Acceptability of Intervention Measure (AIM) Score | 6 and 12 months
  Satisfaction with implementation package will be measured by the 4-item validated Acceptability of Intervention Measure. Mean scores between 1 and 5 will be reported, where higher scores increased acceptability.
Intervention Appropriateness Measure (IAM) Score | 6 and 12 months
  Fit and relevance of the implementation package will be measured by the 4-item validated Intervention Appropriateness Measure. Mean scores between 1 and 5 will be reported, where higher scores increased appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Julia R Berian, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, by request only with IRB approval
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after study completion
Access Criteria: Deidentified, by request only with IRB approval

REFERENCES:
- [Background] Eamer G, Taheri A, Chen SS, Daviduck Q, Chambers T, Shi X, Khadaroo RG. Comprehensive geriatric assessment for older people admitted to a surgical service. Cochrane Database Syst Rev. 2018 Jan 31;1(1):CD012485. doi: 10.1002/14651858.CD012485.pub2. PMID 29385235
- [Background] McDonald SR, Heflin MT, Whitson HE, Dalton TO, Lidsky ME, Liu P, Poer CM, Sloane R, Thacker JK, White HK, Yanamadala M, Lagoo-Deenadayalan SA. Association of Integrated Care Coordination With Postsurgical Outcomes in High-Risk Older Adults: The Perioperative Optimization of Senior Health (POSH) Initiative. JAMA Surg. 2018 May 1;153(5):454-462. doi: 10.1001/jamasurg.2017.5513. PMID 29299599
- [Background] Partridge JS, Harari D, Martin FC, Peacock JL, Bell R, Mohammed A, Dhesi JK. Randomized clinical trial of comprehensive geriatric assessment and optimization in vascular surgery. Br J Surg. 2017 May;104(6):679-687. doi: 10.1002/bjs.10459. Epub 2017 Feb 15. PMID 28198997
- [Background] Chow WB, Rosenthal RA, Merkow RP, Ko CY, Esnaola NF; American College of Surgeons National Surgical Quality Improvement Program; American Geriatrics Society. Optimal preoperative assessment of the geriatric surgical patient: a best practices guideline from the American College of Surgeons National Surgical Quality Improvement Program and the American Geriatrics Society. J Am Coll Surg. 2012 Oct;215(4):453-66. doi: 10.1016/j.jamcollsurg.2012.06.017. Epub 2012 Aug 21. No abstract available. PMID 22917646